CLINICAL TRIAL: NCT03711526
Title: Prognostic Value of Preoperative 6-Minute Walk Test in Patients Undergoing Laparoscopic Gastrointestinal Surgery: a Prospective Cohort Study
Brief Title: Prognostic Value of Preoperative 6-Minute Walk Test for Laparoscopic Gastrointestinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LZJ001
Record Dates: First submitted 2018-10-10; First posted 2018-10-18 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-05

CONDITIONS: Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
6-minute walk test (6MWT) is widely used in cardiopulmonary surgery as a prognostic marker. This prospective cohort study aims to find whether 6MWT will be a good prognostic factor for patients who will undergo laparoscopic gastrointestinal surgery.The investigators will enroll patients awaiting elective laparoscopic gastrointestinal surgery in this study. After informed consent was obtained, the participants will be evaluated through 6MWT. Preoperative assessment and conditions during operation will be recorded. The investigators will analyze the correlation between preoperative 6MWT's result and outcomes after laparoscopic gastrointestinal surgery.

DETAILED DESCRIPTION:
This is a prospective observational cohort study, which focus on the prognostic value of 6-minute walk test (6MWT) in patients who will undergo laparoscopic gastrointestinal surgery.

Enhanced recovery after surgery (ERAS) is an optimized program which help patients accelerate recovery and improve outcomes by integrating evidence-based protocols and guidelines. With the rapid development of ERAS, the preoperative clinical data of patients are paid more and more attention to evaluate the risk of perioperative complications and choose an appropriate time for surgery. A better perioperative evaluation method will lead to lower morbidity and mortality rates of postoperative complications and shorter time of hospital stay. So, it is important to find an appropriate evaluation method to predict the outcomes of patients undergoing surgery.

6MWT is a low-cost, easy to operate and well-tolerated test to evaluate exercise tolerance to predict cardiopulmonary function. It has widely used in cardiopulmonary surgery as a prognostic marker. Even though massive studies showed that decreased perioperative 6-minute walk distance (6MWD) related to postoperative complication in patients underwent cardiac or pulmonary surgery, there are only small numbers of studies with small number sizes presenting correlation of decreased 6MWD and postoperative complication in abdominal surgery. Even some studies of upper abdomen got the opposite result. Furthermore, the critical value for 6MWD is still controversial. Based on these conditions, this study was designed to investigate if 6MWT cloud be used as an accurate assessment with the prognostic value in patients who will undergo laparoscopic gastrointestinal surgery to improve the ERAS program.

The investigators decide to enroll 200 patients awaiting elective laparoscopic gastrointestinal surgery in this study at Peking Union Medical College Hospital. After informed consent was obtained, the patients will be comprehensively evaluated from demographic characteristics, complications of systems and organs, laboratory tests results, 6MWT, metabolic equivalents (METs), psychological states assessed by hospital anxiety and depression scale. Outcomes will be assessed according to the Clavien-Dindo Classification of Surgical Complications. Operative name, operation date, operative method, blood loss, situation of blood transfusion, operation time, duration of anesthesia, whether return to ICU or not (treatment time and tubulization time), drainage flow of within 24 hours after surgery will be recorded. Other outcome measures include the mortality rate within 30 days after surgery, second operation without plan, rehospitalized rate without plan, postoperative hospitalization time, patient satisfaction.

Descriptive analysis, univariate analysis, multivariate analysis and establishment of complication prediction model will be used to analyze the correlation between preoperative 6MWD and outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatient in Peking Union Medical College Hospital from January 2019 to December 2019
2. From 18 y/o to 75 y/o
3. Consent got from patients
4. Decide to take the elective laparoscopic gastrointestinal surgery in Peking Union Medical College Hospital

Exclusion Criteria:

1. Refuse to take part in the study (due to any reason)
2. ASA grade ≥ IV
3. Unable to cooperate with the study (mental disorder, disturbance of consciousness, dysnoesia)
4. Have developed unstable angina or myocardial infarction in the recent 6 months
5. HR>120 beats/min or SBP>180mm/Hg or DBP>100mmHg at resting state
6. During acute episode of asthma
7. Diseases cause severe limitation of walking, including severe lumbar spondylosis, knee osteoarthritis, lower extremity varicose veins, et al.
8. Other conditions make patients can't cooperate with 6MWT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inpatient from 18 y/o to 75 y/o going to have elective laparoscopic gastrointestinal surgery in Peking Union Medical College Hospital from January 2019 to December 2019.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  Postoperative complications includes postoperative wound infections, delayed union or nonunion, intraperitoneal abscesses, intestinal obstruction, anastomotic fistula, postoperative hemorrhage which need blood transfusion, pulmonary complications, cardiovascular complications, cerebrovascular complications, thrombotic events, acute liver failure or deterioration of liver function, acute renal failure or deterioration of renal function, urinary infection, gastrointestinal hemorrhage, postoperative delirium, et al.

SECONDARY OUTCOMES:
Mortality rate | 30 days
  Postoperative death due to any reason
Second operation without plan | 30 days after surgery
  During the same hospital stay, unplanned reoperations were performed for a variety of reasons.
Rehospitalized | 30 days
  Rehospitalized without plan due to any reason
Patient satisfaction | 30 days
  telephone visits by a blinded doctor with same standardized questions were conducted.

CONTACTS AND LOCATIONS:
Overall Officials: YUGUANG HUANG, MD., Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Y, Liu Z, Zhang L, Zhang Y, Zhang N, Han Y, Shen L. Preoperative 6-minute walk distance is associated with postoperative complications in patients undergoing laparoscopic gastrointestinal cancer surgery. Eur J Surg Oncol. 2024 Jan;50(1):107139. doi: 10.1016/j.ejso.2023.107139. Epub 2023 Nov 4. PMID 37948791